CLINICAL TRIAL: NCT00004163
Title: Herceptin In Patients With Advanced or Metastatic Salivary Gland Carcinomas
Brief Title: Trastuzumab in Treating Patients With Advanced Salivary Gland Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Robert I. Haddad, MD, Haddad, Robert MD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 98-286; P30CA006516 (NIH); NCI-G99-1628; CDR0000067405 (Other: Other)
Record Dates: First submitted 1999-12-10; First posted 2004-03-15 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Head and Neck Cancer
Keywords: stage III salivary gland cancer; stage IV salivary gland cancer; recurrent salivary gland cancer; salivary gland squamous cell carcinoma; salivary gland acinic cell tumor; low-grade salivary gland mucoepidermoid carcinoma; high-grade salivary gland mucoepidermoid carcinoma; salivary gland adenocarcinoma; salivary gland poorly differentiated carcinoma; salivary gland malignant mixed cell type tumor; salivary gland adenoid cystic carcinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Salivary Gland Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Trastuzumab (Experimental): * Trastuzumab is administered intravenously weekly
  * CAT or MRI scans will be performed every 2 cycles
  Interventions: Drug: Trastuzumab

INTERVENTIONS:
Drug: Trastuzumab
  Other Names: Herceptin

SUMMARY:
RATIONALE: Monoclonal antibodies, such as trastuzumab, can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase II trial to study the effectiveness of trastuzumab in treating patients who have advanced salivary gland cancer.

DETAILED DESCRIPTION:
Due to the age of this study upon transfer from the NCI to DFCI, data was not accessible to find the exact primary completion date (PCD) or study completion date (SCD). The September 2001 date used for both is based on known enrollment dates and an estimate on median time to progression (TTP) in the setting of this clinical trial. Since participants were treated indefinitely until progression, TTP is deemed to reflect generally the time on treatment for evaluation of the primary response outcome. Furthermore, patients were followed for progression to estimate TTP, a secondary outcome measure.

OBJECTIVES: I. Determine the response rate to trastuzumab in patients with advanced or metastatic salivary gland cancer. II. Determine the time to progression in these patients after this regimen. III. Determine the toxicity of trastuzumab in these patients.

OUTLINE: Patients are stratified according to histology: intercalated duct (adenoid cystic carcinoma, acinic cell carcinoma, malignant mixed tumor, polymorphous low grade adenocarcinoma, undifferentiated carcinoma, adenocarcinoma) vs excretory duct (squamous cell carcinoma, mucoepidermoid carcinoma).

PROJECTED ACCRUAL: A total of 50 patients (25 per stratum) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria

* Histologic diagnosis of any of the following malignancies originating from salivary tissue: adenoid cystic carcinoma, mucoepidermoid carcinoma, acinic cell carcinoma, malignant mixed tumor, polymorphous low grade adenocarcinoma, undifferentiated carcinoma, squamous cell carcinoma, adenocarcinoma.
* Her2/neu determination: Patients must have overexpression of the Her2/neu protein in the tumor documented by the Dako polyclonal rabbit anti-Her2 antisera assay.

Overexpression may be documented by staining of the original paraffin embedded tumor from the time of diagnosis or from material obtained at the time of locoregional or distant recurrence.

Overexpression of HER2/neu will be per the Dako Herceptest guidelines. A Score of 2+ or 3+ will be defined as overexpression. All slides will be reviewed by members of the departments of pathology at either the Brigham and Women's Hospital or the Beth Israel Hospital in Boston.

* Patients must be incurable on the basis of unresectable local or distant disease as determined by the patient's surgeon.
* Patients must have an ECOG performance status of 0 to 1.
* Patients must have at least uni-dimensionally measurable disease documented within one month of initiation of treatment. Measurement may be by physical exam or radiologically. Attempts should be made to photo document all tumor sites assessed by physical examination with a metric ruler within the photo for measurement confirmation.
* Patients must be willing and able to go through the process of informed consent.
* Patients must have a life expectancy exceeding 3 months.
* Patients must be at least 18 years old.
* Patients must have adequate organ function as defined by the following tests to be performed within 14 days of therapy initiation:

  * Absolute neutrophil count > 1999 cells x 10 61L
  * Platelet count > 99,999 cells x 106/L
  * Hemoglobin >8.5 gm/di or HCT > 25%
  * Serum creatinine < 1.5 x institutional upper limits of normal (ULN) or creatinine clearance measured by 24 hour urine collection as at least 50% of institutional lower limit of normal.
  * Total bilirubin <2 x institutional ULN
  * AST (SGOT) < 2 x institutional ULN *
* If from documented liver involvement with cancer, may be up to < 5 x institutional ULN Alkaline Phosphatase < 5 x institutional ULN *
* If from documented bone or liver involvement with cancer, no upper limit restriction.
* Baseline determination of normal left ventricular ejection fraction as evidenced MUGA or echocardiogram.

Exclusion Criteria:

* Patients must not have received more than two regimens of cytotoxic chemotherapy for salivary gland cancer. Previous immunologic, hormonal, homeopathic, natural, or alternative medicine therapies are acceptable provided treatment ended greater than 28 days prior to protocol therapy.
* Patients must not receive any form (including radiotherapeutic, immunologic, hormonal, homeopathic, natural, or alternative medicine) of anti-neoplastic therapy other than Herceptin while participating in this study.
* Patients must not have a history of any non-salivary invasive neoplasm within three years of trial entry, excepting curatively treated non-melanoma skin cancer and cervical cancer.
* Pregnant and breast feeding women are not eligible for this study. No pregnancy test is required. Women of childbearing potential must be counseled on the use of effective birth control prior to participation in this study.
* Patients with significant active illness (e.g. congestive heart failure, COPD, uncontrolled diabetes, AIDS, previous MI, cardiomyopathies, history of uncontrolled arrhythmias) are not eligible for this study.
* Patients who have received anthracyclines (e.g. doxorubicin, daunorubicin, epirubicin) are eligible but must have a baseline MUGA scan documenting normal cardiac contractility (at or above the normal institutional limit) within one month of trial enrollment. The upper limit of doxorubicin exposure should be no more than 360mg1m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1999-10 (Actual); Primary Completion 2001-09 (Actual); Study Completion 2001-09 (Actual)

PRIMARY OUTCOMES:
Response Rate | 2 years

SECONDARY OUTCOMES:
Time to Progression | 2 years
Toxicity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Marshall R. Posner, MD, Study Chair — Dana-Farber Cancer Institute
Locations (10):
- United States (10):
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Hematology/Oncology Associates, Port Saint Lucie, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Cape Cod Health Care, Hyannis, Massachusetts
  - Nantucket Cottage Hospital, Nantucket, Massachusetts
  - Washington University Barnard Cancer Center, St Louis, Missouri
  - Lourdes Regional Cancer Center, Binghamton, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No